CLINICAL TRIAL: NCT02766270
Title: A Prospective Study of Concurrent Chemoradiotherapy With Temozolomide Versus Radiation Therapy Alone in Patients With IDH Wild-type/TERT Promoter Mutation Grade II/III Gliomas
Brief Title: CCRT With Temozolomide Versus RT Alone in Patients With IDH Wild-type/TERT Promoter Mutation Grade II/III Gliomas
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Tao Jiang, Vice Director of Neurosurgical Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFMD 2016-2-1073
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Grade II/III Glioma
Keywords: Grade II/III Glioma; IDH; TERT; Chemoradiotherapy; Temozolomide
MeSH Terms: interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiotherapy with Temozolomide (Experimental): Patients undergo intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy 5 days a week for 6 weeks (for a total of 60 Gy) and receive temozolomide PO QD (75 mg/m2/day, 7 days/week) for up to 7 weeks. Beginning 4 weeks after completion of chemotherapy and radiation therapy, patients receive temozolomide PO QD on days 1-5 (150-200 mg/m2). Treatment with temozolomide repeats every 28 days for up to 12 courses
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy
- Radiotherapy alone (Active Comparator): Patients undergo intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy 5 days a week for 6 weeks (for a total of 60 Gy)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Temozolomide — RT with daily temozolomide (75 mg/m2/day, 7 days/week for up to 7 weeks) and adjuvant temozolomide (150-200 mg/m2 PO QD for 5 days, repeats every 28 days for up to 12 courses).
  Arms: Chemoradiotherapy with Temozolomide
Radiation: Radiotherapy

SUMMARY:
The management of lower-grade gliomas (Diffuse low-grade and intermediate-grade gliomas, WHO II and III) is largely based on surgery followed by radiotherapy. Recent studies showed that lower-grade glioma patients with IDH wild-type (IDH-wt) and TERT promoter mutation (TERTp-mut) had dismal clinical outcomes. These results suggested that current treatment strategies are not adequate for this subtype of lower-grade glioma.

The present study aims to examine the efficacy and safety of concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide for lower- grade glioma patients with IDH-wt and TERTp-mut.

DETAILED DESCRIPTION:
Diffuse low-grade and intermediate-grade gliomas (which together make up the lower-grade gliomas, World Health Organization grades II and III) are infiltrative neoplasms that arise most often in the cerebral hemispheres of adults and include astrocytomas, oligodendrogliomas, and oligoastrocytomas. The management of lower-grade gliomas is largely based on surgery followed by radiotherapy.

Lower-grade gliomas have highly variable clinical behavior that is not adequately predicted on the basis of histologic class. Consequently, clinicians increasingly rely on genetic classification to guide clinical decision making. Mutations in IDH1 and IDH2 characterize the majority of lower-grade gliomas in adults and define a subtype that is associated with a favorable prognosis. Mutations of the telomerase reverse transcriptase (TERT) promoter, which result in enhanced telomerase activity and lengthened telomeres, have been observed in several human cancers including glioma. Accumulating evidence suggest that TERT promoter mutation is another molecular marker which can stratify lower-grade gliomas into prognostic subgroups in combination with IDH mutation. In our previous study, patients(28/377, 7.4%) who had lower-grade gliomas with IDH wild-type (IDH-wt) and TERT promoter mutation (TERTp-mut) had the poorest clinical outcomes (median OS, 27.7mo; 5-year OS, 29%). These results were accordant with the recent studies and suggested that current treatment strategies are not adequate for this subtype of lower-grade glioma.

Radiotherapy plus temozolomide has emerged as a new standard of care for patients with good PS non-elderly glioblastoma. There are some data that support temozolomide as adjuvant therapy for lower-grade glioma. Given that the IDH-wt/TERTp-mut subgroup of lower-grade gliomas has dismal prognosis, a more aggressive therapy such as concurrent chemoradiotherapy seems to be reasonable. The present study aims to examine the efficacy and safety of concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide for lower-grade glioma patients with IDH-wt and TERTp-mut. Half the patients will be randomly assigned to receive concurrent chemoradiotherapy (surgery + concurrent chemoradiotherapy with temozolomide followed by adjuvant temozolomide) and half the patients will be randomly assigned to receive conventional therapy (surgery + radiotherapy only).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial Diffuse low-grade and intermediate-grade gliomas (World Health Organization grades II and III )
* IDH wild-type and TERT promoter mutation
* Age > 18
* Karnofsky performance score > 60
* Neutrophilic granulocyte count > 1500/µl
* Platelet count > 100 000/µl
* Hemoglobin > 10 g/dl
* Serum creatinine < 1.5 times the lab's upper normal limit
* AST or ALT < 1.5 times the lab's upper normal limit
* Adequate medical health to participate in this study
* No previous systemic chemotherapy
* No previous radiotherapy to the brain
* Written informed consent

Exclusion Criteria:

* Serious medical or neurological condition with a poor prognosis
* Contraindications to radiotherapy or temozolomide chemotherapy
* Patient unable to follow procedures, visits, examinations described in the study
* Second cancer requiring radiotherapy or chemotherapy
* Inability to undergo gadolinium-contrasted MRIs
* Pregnant women or nursing mothers can not participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from randomization to death.

SECONDARY OUTCOMES:
Progression free survival(PFS) | Up to 2 years
  Progression free survival(PFS) is defined as the time from randomization to progressive disease or death. A combination of neurological examination and MRI brain scan used to define progression.
The incidence and severity of adverse events associated with treatment with RT alone and combined with temozolomide chemotherapy; according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan H, Parsons DW, Jin G, McLendon R, Rasheed BA, Yuan W, Kos I, Batinic-Haberle I, Jones S, Riggins GJ, Friedman H, Friedman A, Reardon D, Herndon J, Kinzler KW, Velculescu VE, Vogelstein B, Bigner DD. IDH1 and IDH2 mutations in gliomas. N Engl J Med. 2009 Feb 19;360(8):765-73. doi: 10.1056/NEJMoa0808710. PMID 19228619
- [Background] Parsons DW, Jones S, Zhang X, Lin JC, Leary RJ, Angenendt P, Mankoo P, Carter H, Siu IM, Gallia GL, Olivi A, McLendon R, Rasheed BA, Keir S, Nikolskaya T, Nikolsky Y, Busam DA, Tekleab H, Diaz LA Jr, Hartigan J, Smith DR, Strausberg RL, Marie SK, Shinjo SM, Yan H, Riggins GJ, Bigner DD, Karchin R, Papadopoulos N, Parmigiani G, Vogelstein B, Velculescu VE, Kinzler KW. An integrated genomic analysis of human glioblastoma multiforme. Science. 2008 Sep 26;321(5897):1807-12. doi: 10.1126/science.1164382. Epub 2008 Sep 4. PMID 18772396
- [Background] Killela PJ, Reitman ZJ, Jiao Y, Bettegowda C, Agrawal N, Diaz LA Jr, Friedman AH, Friedman H, Gallia GL, Giovanella BC, Grollman AP, He TC, He Y, Hruban RH, Jallo GI, Mandahl N, Meeker AK, Mertens F, Netto GJ, Rasheed BA, Riggins GJ, Rosenquist TA, Schiffman M, Shih IeM, Theodorescu D, Torbenson MS, Velculescu VE, Wang TL, Wentzensen N, Wood LD, Zhang M, McLendon RE, Bigner DD, Kinzler KW, Vogelstein B, Papadopoulos N, Yan H. TERT promoter mutations occur frequently in gliomas and a subset of tumors derived from cells with low rates of self-renewal. Proc Natl Acad Sci U S A. 2013 Apr 9;110(15):6021-6. doi: 10.1073/pnas.1303607110. Epub 2013 Mar 25. PMID 23530248
- [Background] Nonoguchi N, Ohta T, Oh JE, Kim YH, Kleihues P, Ohgaki H. TERT promoter mutations in primary and secondary glioblastomas. Acta Neuropathol. 2013 Dec;126(6):931-7. doi: 10.1007/s00401-013-1163-0. Epub 2013 Aug 17. PMID 23955565
- [Background] Yang P, Cai J, Yan W, Zhang W, Wang Y, Chen B, Li G, Li S, Wu C, Yao K, Li W, Peng X, You Y, Chen L, Jiang C, Qiu X, Jiang T; CGGA project. Classification based on mutations of TERT promoter and IDH characterizes subtypes in grade II/III gliomas. Neuro Oncol. 2016 Aug;18(8):1099-108. doi: 10.1093/neuonc/now021. Epub 2016 Mar 7. PMID 26957363
- [Background] Chan AK, Yao Y, Zhang Z, Chung NY, Liu JS, Li KK, Shi Z, Chan DT, Poon WS, Zhou L, Ng HK. TERT promoter mutations contribute to subset prognostication of lower-grade gliomas. Mod Pathol. 2015 Feb;28(2):177-86. doi: 10.1038/modpathol.2014.94. Epub 2014 Aug 1. PMID 25081751
- [Background] Labussiere M, Di Stefano AL, Gleize V, Boisselier B, Giry M, Mangesius S, Bruno A, Paterra R, Marie Y, Rahimian A, Finocchiaro G, Houlston RS, Hoang-Xuan K, Idbaih A, Delattre JY, Mokhtari K, Sanson M. TERT promoter mutations in gliomas, genetic associations and clinico-pathological correlations. Br J Cancer. 2014 Nov 11;111(10):2024-32. doi: 10.1038/bjc.2014.538. Epub 2014 Oct 14. PMID 25314060
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Quinn JA, Reardon DA, Friedman AH, Rich JN, Sampson JH, Provenzale JM, McLendon RE, Gururangan S, Bigner DD, Herndon JE 2nd, Avgeropoulos N, Finlay J, Tourt-Uhlig S, Affronti ML, Evans B, Stafford-Fox V, Zaknoen S, Friedman HS. Phase II trial of temozolomide in patients with progressive low-grade glioma. J Clin Oncol. 2003 Feb 15;21(4):646-51. doi: 10.1200/JCO.2003.01.009. PMID 12586801
- [Derived] Zhang J, Wang P, Ren Y, Chen L, Feng J, Liu F, Deng K, Bao Z, Qiu X, Liu Y. Chemoradiotherapy with temozolomide vs. radiotherapy alone in patients with IDH wild-type and TERT promoter mutation histological grade 2/3 gliomas: An extension retrospective analysis of a randomized controlled trial. Cancer. 2025 Dec 1;131(23):e70171. doi: 10.1002/cncr.70171. PMID 41328764
- [Derived] Qiu X, Chen Y, Bao Z, Chen L, Jiang T. Chemoradiotherapy with temozolomide vs. radiotherapy alone in patients with IDH wild-type and TERT promoter mutation WHO grade II/III gliomas: A prospective randomized study. Radiother Oncol. 2022 Feb;167:1-6. doi: 10.1016/j.radonc.2021.12.009. Epub 2021 Dec 10. PMID 34902368